CLINICAL TRIAL: NCT07374809
Title: DISSECTING THE EPIGENOME AND MICROENVIRONMENT TO UNDERSTAND IMMUNOTHERAPY EFFICACY TARGETING ENDOMETRIAL CANCER (DEMETER PROJECT)
Brief Title: IMMUNOTHERAPY EFFICACY TARGETING ENDOMETRIAL CANCER
Acronym: DEMETER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UID 5032; L2-516 (Other: Comitato Etico Territoriale Lombardia 2)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Carcinoma (EC); pMMR; DMMR Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm 1 (Experimental): Histologically confirmed epithelial endometrial carcinoma (endometrioid, serous, clear cell, mixed histology, or carcinosarcoma), classified as dMMR or pMMR -Availability of a fresh tumor sample suitable for study procedures
  Interventions: Diagnostic Test: DNA methylation profiles

INTERVENTIONS:
Diagnostic Test: DNA methylation profiles — MAP mutations, DNA methylation profiles, transcriptome, TME composition, and lipid abundance of tumor samples from EC patients that underwent immunotherapy;

SUMMARY:
Endometrial carcinoma (EC) represents the most common gynecological malignancy in developed countries. Despite therapeutic advances, patients with advanced or recurrent disease still have a poor prognosis, with high recurrence rates and a 5-year survival of less than 20%.

Recently, four phase III studies (RUBY, NRG-GY018, AtTEnd, and DUO-E) have demonstrated that the addition of anti-PD-1/PD-L1 immunotherapy to first-line chemotherapy significantly improves progression-free survival, particularly in tumors with altered DNA repair mechanisms known as mismatch repair (MMR) (so-called mismatch repair-deficient or dMMR tumors), but with benefits also observed in a subset of tumors with normal MMR function (so-called MMR-proficient or pMMR tumors). However, despite the clinical approval of these therapies, reliable biomarkers capable of predicting response to immunotherapy are still lacking.

This project aims to comprehensively characterize the genomic, epigenetic, and lipid properties of the tumor and the tumor microenvironment (TME) in order to identify predictive markers of response to immunotherapy, thereby laying the foundation for a personalized therapeutic approach in endometrial carcinoma.

DETAILED DESCRIPTION:
Primary objective To identify and validate predictive biomarkers of response to immunotherapy in dMMR and pMMR endometrial carcinomas through an integrated multi-omics approach (genomic, epigenomic, transcriptomic, and lipidomic) and functional validation in patient-derived models.

Population characteristics Patients with advanced (stage III-IV) or recurrent epithelial endometrial carcinoma, treated with anti-PD-1/PD-L1 immunotherapy in combination with or following standard platinum-based chemotherapy at the European Institute of Oncology.

Inclusion criteria:

Advanced or recurrent endometrial carcinoma patients undergoing biopsy or cytoreductive surgery followed by immunotherapy

Age ≥ 18 years

Fresh tumor tissue available at the IEO Biobank

Written informed consent

Exclusion criteria:

Mesenchymal tumors

Carcinomas of non-endometrial origin

Chronic viral infections (HIV, HBV, HCV)

Number of patients and main criteria

* Total number of planned patients: 50
* Number of IEO patients: 50
* Competitive: No
* Special population: Rare disease / advanced tumor
* Sex and menopausal status: Female, pre- or post-menopausal
* Disease stage: III-IV (advanced or recurrent)
* Main subtypes: dMMR and pMMR; molecular subgroups (POLE, p53, NSMP) when available

Duration (in months)

* Enrollment duration: 18
* Follow-up duration: 12 (calculated from the last patient enrolled)

Rationale: with approximately 150 new EC cases per year at IEO (about 20% advanced/recurrent), enrolling 50 patients over 18 months is realistic; a 12-month follow-up allows for clinical evaluations (response/early PFS) that are useful for multi-omics analyses and validation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years old.
* Histologically confirmed epithelial endometrial carcinoma (endometrioid, serous, clear cell, mixed, or carcinosarcoma).
* Advanced (stage III-IV) or recurrent disease, eligible for surgery or biopsy as part of the therapeutic plan.
* Availability of fresh-frozen or OCT-embedded tumor tissue obtained at surgery/biopsy and stored in the IEO Biobank.
* Mismatch-repair-deficient (dMMR) or -proficient (pMMR) molecular subtype (when available).
* Written informed consent for participation and use of biological material for translational research purposes.

Exclusion Criteria:

* Mesenchymal tumors or epithelial tumors of non-endometrial origin (e.g., ovarian, cervical).
* Prior systemic treatment with immune checkpoint inhibitors for other malignancies.
* Insufficient or poor-quality tumor tissue available for molecular analyses.
* Active or uncontrolled infection with HIV, HBV, or HCV.
* Any condition that, in the investigator's judgment, would compromise patient safety or study integrity.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
predictive biomarkers | 2 years
  To identify and validate predictive biomarkers of response to immunotherapy in dMMR and pMMR endometrial carcinomas through an integrated multi-omics approach (genomic, epigenomic, transcriptomic, and lipidomic) and functional validation in patient-derived models.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Europeo di Oncologa, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No